CLINICAL TRIAL: NCT05864976
Title: Advancing Neurosurgical Neuronavigation Using Resting State MRI and Machine Learning - a Prospective Study
Brief Title: Neurosurgical Neuronavigation Using Resting State MRI and Machine Learning
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 202305045; 2R01CA203861 (NIH)
Record Dates: First submitted 2023-05-08; First posted 2023-05-18 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Standard of care rsfMRI using the Support Vector Machine algorithm: * Once enrolled, clinical pre-surgical MRI will be done on Siemens 3T Prisma or Skyra scanners using a standard pre-surgical tumor protocol. Resting-state functional MRI (rsfMRI) will be acquired. The Support Vector Machine (SVM) algorithm will be used on this pre-surgical MRI.
  * Patients will undergo post-operative MRI at approximately 8-12 weeks following surgical resection to evaluate extent of resection. Patients will then undergo subsequent MRI imaging every 2-3 months as part of routine clinical care to monitor for recurrence. The following MR sequences will be acquired: pre-and post-contrast T1-weighted, T2-weighted FLAIR, diffusion weighted imaging. MRI scans will be reviewed by a board-certified neuroradiologist to determine date of radiographic progression/recurrence. Imaging features at recurrence including location, multifocality, and presence of diffuse or distant recurrence will also be recorded.
  Interventions: Device: Support Vector Machine

INTERVENTIONS:
Device: Support Vector Machine — Machine learning algorithm

SUMMARY:
This study is investigating the use of a computer algorithm to analyze scans of the brain before surgery to predict how a person's tumor will respond to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Must have a radiological diagnosis of a lesion in the brain with characteristics consistent with glioblastoma multiforme.
* Must be planning to undergo a pre-operative MRI.
* Must be at least 18 years old.
* Must be able to understand and willing to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Contraindication to MRI.
* Inability to have clinical follow-up (e.g., patient is out of town and will do follow-up elsewhere).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants being seen at Washington University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-06 (Actual); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants who are deemed as short-term survivor or a long-term survivor | Through completion of follow-up (estimated to be 2 years)
  -Patients will be deemed as a short-term survivor or a long-term survivor and this will be defined as overall survival as less than or greater than 14.5 months, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Mathios, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu